CLINICAL TRIAL: NCT06078449
Title: Effect of Ultrasound With Simultaneous Hyaluronate Injection on Risk of Fall in Geriatric Women With Knee Osteoarthritis
Brief Title: Ultrasound Effect With Hyaluronate Injection on Risk of Fall in Geriatric Women With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Hend Reda Sakr, Lecturer of Physical Therapy for Woman's Health, Badr University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hend 5
Record Dates: First submitted 2023-02-08; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Osteo Arthritis Knee
Keywords: Risk of fall; osteoarthritis; hyaluronate; geriatric females
MeSH Terms: conditions — Osteoarthritis | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection group (Experimental): Group (1) the study group, they will receive HA intra-articular injection in addition to 12 sessions of therapeutic ultrasound.
  Interventions: Device: Therapeutic Ultrasonic; Drug: Hyaluronan intra-articular injection
- Ultrasound group (Other): Group (2) served as the control group, will receive only HA intra-articular knee injection.
  Interventions: Drug: Hyaluronan intra-articular injection

INTERVENTIONS:
Device: Therapeutic Ultrasonic — Ultrasound is a therapeutic modality that has been used by physical therapists to achieve therapeutic benefits. It is alternating compression and rarefaction of sound waves with a frequency of >20,000 cycles/second. Therapeutic ultrasound frequency will be used by 0.7 to 3.3 MHz. Maximum energy absorption in soft tissue will be 2 to 5 cm. Intensity decreases as the waves penetrate deeper. It is applied using a round headed wand or probe that is put in direct contact with the patient's skin. Ultrasound gel must be used on all surfaces of the head as a conducting medium in order to assist in the transmission of the ultrasonic waves & to reduce friction.
  Arms: Injection group
Drug: Hyaluronan intra-articular injection — The type of Hyaluronan injection that will be used in this study consists of High Molecular Weight Hyaluronic acid (High MW HA 3000 kDa), will be given by the orthopedic surgeon.

SUMMARY:
For many years' physiotherapists have been using ultrasound in treatment of knee osteoarthritis especially in geriatrics (people aged above 65 years) for its known therapeutic effect in relieving pain and improving knee function. Hyaluronan is used to treat osteoarthritis of the knee. Such treatments, called viscosupplementation, are administered as a course of injections into the knee joint, and are believed to supplement the viscosity of the joint fluid, thereby lubricating the joint, cushioning the joint, and producing an analgesic effect. Studies reveals the risk for falls increases with additional symptomatic OA lower limb joints and confirms in addition to gender factor; including female sex.

DETAILED DESCRIPTION:
It is hypothesized that physical therapy by ultrasound might add some extra benefit on risk of fall when applied after intra-articular hyaluronate of Knee OA in female geriatrics. So, forty female geriatrics with ages ranged from 65 to 75 years, randomly will be selected from Ahmed Maher Teaching Hospital, Kasr el einy hospital, Charity clinic and Outpatient clinic of Badr university, referred to physical therapy by an orthopedic surgeon. All will be diagnosed as chronic OA of one or both knees where conventional therapeutic measures failed. They will be assigned to begin HA intra-articular knee injection by the orthopedic surgeon once weekly for 3 weeks. These patients will be randomly divided into 2 groups equal in number, group (1) the study group, they will receive HA intra-articular injection in addition to 12 sessions of therapeutic ultrasound, while group (2) served as the control group receiving only HA intra-articular knee injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients' ages above 65 years.
* Patients diagnosed as chronic osteoarthritis of more than 5 years.
* The OA diagnosed as grade (III to V)
* Patients failed with conventional treatment.
* All patients followed up with the same orthopedic surgeon, and they took the same type of HA intra-articular injection (HA of High MW 3000 kDa).
* All patients were medically stable and do not suffer from any other diseases which may affect the trial results.
* All patients were not treated with analgesics or any medication which may cause misleading results.
* None of the patients received intra-articular hyaluronic acid injection for 1 year or intra-articular corticosteroid injection within the last 3 months.
* All patients didn't take or oral glucosamine or chondroitin supplements or stopped these drugs 2-3 months before participating in this study.
* Every patient signed a consent form.

Exclusion Criteria:

* Young individuals (their age is below 65 years old).
* Mild degree of OA (grade I & II).
* Patients who had undergone knee arthroscopy, or any knee surgery.
* Patients with OA secondary to trauma.
* Patients with metal implants.
* Patients with CNS dysfunction.

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Females are affected more than males due to menopausal changes and declined estrogen hormone that accelerates bone loss and leads to high risk of fall and decreased balance due to orthopedic issues.
Enrollment: 40 (Estimated)
Dates: Start 2023-11-11 (Estimated); Primary Completion 2024-03-11 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
ROM | At the beginning of study, we measure range of motion in patients in both groups then after one month to assess progression of range of motion in both groups.
  Range of motion by using OB Goniometer "Myrin"
6 min walk test | At the beginning of study, we assess balance by 6 min walk test in patients in both groups then after one month to assess progression in balance in both groups.
  The 6MWT required a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measured the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
Berg balance scale | At the beginning of study, we assess balance by Berg balance scale in patients in both groups then after one month to assess progression in balance in both groups.
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Badr University, Cairo, New Cairo, Egypt